CLINICAL TRIAL: NCT01240889
Title: Effects of Intranasal Corticosteroid and Montelukast On Nasal Allergen Challenges*
Acronym: Roche
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Thomas B. Casasle, MD, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-15912
Record Dates: First submitted 2010-10-28; First posted 2010-11-15 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Allergy
Keywords: Ragweed allergies; acoustic rhinometry; nasal allergen challenge
MeSH Terms: conditions — Hypersensitivity | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- montelukast (Active Comparator): luekotriene inhibitor
  Interventions: Drug: Fluticasone
- Fluticasone (Active Comparator): Nasal steroid
  Interventions: Drug: Fluticason

INTERVENTIONS:
Drug: Fluticasone — nasal spray
  Arms: montelukast
Drug: Fluticason — 2 sprays per day in each nostril
  Arms: Fluticasone

SUMMARY:
This study will be a randomized, double blind, placebo-controlled, parallel group study and will include subjects with ragweed-induced seasonal allergic rhinitis.

DETAILED DESCRIPTION:
The primary goal of this proposal is to assess the ability of an intranasal corticosteroid, fluticasone, and montelukast to affect the upper airway and systemic physiologic, biologic and clinical parameters occurring after an early and late upper airway allergic response to ragweed in ragweed allergic rhiniticsThe assessment of early allergy responses in the nose has been fairly well established in our laboratory and we will use methods detailed in previous publications (21, 23 24). One potential challenge will be to sample upper airway mediators and cytokines without affecting clinical parameters such as symptom scores and acoustic rhinometry readings. Moreover, we will need to sample at time points throughout six or more hours in order to accurately determine the effects on late phase allergic responses. Nasal filter paper sampling is a technique that we are currently engaged in using, and we will work with Roche to elute the samples and measure multiple mediators and cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 19-60 years.
* Females of child bearing potential must use appropriate birth control throughout the study and urine pregnancy tests must be negative prior to dosing at each study visit.
* Subjects with a documented history of ragweed-induced seasonal allergic rhinitis requiring pharmacotherapy during the preceding 2 allergen seasons.
* Subjects with a positive skin prick test to short ragweed (Amb a 1) extract, defined as >3mm wheal larger than saline control
* Subjects spirometry FEV1 must be > 80% predicted prior to each allergen challenge
* Subjects average post diluents nasal congestion score must be < 1 at admission for each study visit

Exclusion Criteria:

* Subjects with evidence or history of clinically significant medical illnesses other than changes related to allergic rhinitis. Subjects with some stable chronic medical conditions not expected to interfere with the conduct or safety of the study may be eligible to participate based on the investigator's discretion.
* Subjects with a history of asthma or urticaria, or a screening FEV1 prior to allergen challenge of <80% of predicted. in FEV1 compared to pre-diluent FEV1 baseline at either screening visit.
* Subjects with significant nasal deformity, recent nasal surgery nasal polyps or chronic rhinosinusitis.
* Subjects who have smoked in the last 6 months or have a history of >10 pack years.
* Subjects who are taking or have taken restricted concomitant medications that could confound the safety or efficacy assessments including those shown below.
* Subjects who have history or evidence of alcohol or drug abuse.
* Subjects exposed to cat and have a positive skin test to cat.
* Subjects that have a positive skin test to dust mite (D pteronyssinus/ D farinae) requiring pharmacotherapy

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effect of nasal allergen challenges on biomarkers | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Casale, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513